CLINICAL TRIAL: NCT03469284
Title: Randomized Controlled Trial Comparing 4 Intervention Arms, Including 3 Different Concentrations of Methylene Blue Oral Rinse Combined With Conventional Therapy and Conventional Therapy, in Patients With Intractable Pain Associated With Oral Mucositis
Brief Title: MOM's PAIN (Methylene Blue for Oral Mucositis' PAIN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-1051; NCI-2018-00822 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-1051 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-03-13; First posted 2018-03-19 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Malignant Neoplasm; Oral Pain; Stomatitis
MeSH Terms: conditions — Neoplasms; Stomatitis | interventions — Practice Guidelines as Topic; Standard of Care; Methylene Blue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (lower dose methylene blue, standard of care) (Experimental): Patients receive lower dose methylene blue PO to swish and spit for 5 minutes every 6 hours then receive standard of care therapy.
  Interventions: Other: Best Practice; Drug: Methylene Blue
- Group 2 (medium dose methylene blue, standard of care) (Experimental): Patients receive medium dose methylene blue PO to swish and spit for 5 minutes every 6 hours then receive standard of care therapy.
  Interventions: Other: Best Practice; Drug: Methylene Blue
- Group 3 (higher dose methylene blue, standard of care) (Experimental): Patients receive higher dose methylene blue PO to swish and spit for 5 minutes every 6 hours then receive standard of care therapy.
  Interventions: Other: Best Practice; Drug: Methylene Blue
- Group 4 (standard of care) (Active Comparator): Patients receive standard of care therapy.
  Interventions: Other: Best Practice

INTERVENTIONS:
Other: Best Practice — Given standard of care therapy
  Other Names: standard of care; standard therapy
Drug: Methylene Blue — Given lower dose PO
  Other Names: Azul de Metileno; Azul Metile; Blu di Metilene; CI Basic Blue 9; CI-52015; Collubleu; Colour Index No. 52015; Desmoidpillen; Methylenum Caeruleum; Methylthioninii Chloridum; Methylthioninium Chloride; Schultz No. 1038; Tetramethylthionine Chloride Trihydrate; Urolene Blue; Vitableu
  Arms: Group 1 (lower dose methylene blue, standard of care)
Drug: Methylene Blue — Given medium dose PO
  Other Names: Azul de Metileno; Azul Metile; Blu di Metilene; CI Basic Blue 9; CI-52015; Collubleu; Colour Index No. 52015; Desmoidpillen; Methylenum Caeruleum; Methylthioninii Chloridum; Methylthioninium Chloride; Schultz No. 1038; Tetramethylthionine Chloride Trihydrate; Urolene Blue; Vitableu
  Arms: Group 2 (medium dose methylene blue, standard of care)
Drug: Methylene Blue — Given higher dose PO
  Other Names: Azul de Metileno; Azul Metile; Blu di Metilene; CI Basic Blue 9; CI-52015; Collubleu; Colour Index No. 52015; Desmoidpillen; Methylenum Caeruleum; Methylthioninii Chloridum; Methylthioninium Chloride; Schultz No. 1038; Tetramethylthionine Chloride Trihydrate; Urolene Blue; Vitableu
  Arms: Group 3 (higher dose methylene blue, standard of care)

SUMMARY:
This phase II trial studies how well methylene blue works in treating patients with cancer and pain associated with oral mucositis. Methylene blue may relieve pain associated with oral mucositis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of methylene blue (MB) in reducing the severity of mucositis-related pain, measured by numeric rating scale (NRS), in cancer patients who underwent or are undergoing chemotherapy or radiation therapy.

OUTLINE: Patients are randomized to 1 of 4 groups.

GROUP 1: Patients receive lower dose methylene blue orally (PO) to swish and spit for 5 minutes every 6 hours then receive standard of care therapy.

GROUP 2: Patients receive medium dose methylene blue PO to swish and spit for 5 minutes every 6 hours then receive standard of care therapy.

GROUP 3: Patients receive higher dose methylene blue PO to swish and spit for 5 minutes every 6 hours then receive standard of care therapy.

GROUP 4: Patients receive standard of care therapy.

After completion of study treatment, patients are followed up at 1, 2, 7, and 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cancer diagnosis, receiving chemotherapy, radiation therapy or the combination
* Patients with a current diagnosis of oral mucositis
* Patients with pain and oral dysfunction associated with oral mucositis despite conventional therapy
* Voluntary written consent
* Patient must agree to use of contraception or abstinence from sex during the treatment period and for 30 days after patient's last dose

Exclusion Criteria:

* Patients with known allergy to MB
* Patients taking medications with known significant drug interactions
* Pregnant or lactating patients
* Patients who are cognitively impaired and unable to consent for the study
* Patients with risk of broncho-aspiration based on documented swallowing test by a speech pathologist (if available)
* Patients with known history of G6PD deficiency
* Patients undergoing any other experimental intervention for oral mucositis
* Patients who have no pain or impairment in oral function, patients who are not symptomatic
* Patients with head and neck cancer
* Patients on serotonergic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Roldan, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Roldan CJ, Huh B, Song J, Nieto Y, Osei J, Chai T, Nouri K, Koyyalagunta L, Bruera E. Methylene blue for intractable pain from oral mucositis related to cancer treatment: a randomized phase 2 clinical trial. BMC Med. 2022 Nov 3;20(1):377. doi: 10.1186/s12916-022-02579-8. PMID 36324139
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 1, 2019, and December 01, 2020- Conducted at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: 69 participants signed consent, 9 participants withdrew (3 dropped out of the trial because they were randomized out of the methylene blue group, 5 had progression of disease and could not continue the trial, and 1 was enrolled but withdrew before starting the medication.)
Groups:
- Conventional Therapy (Controlled Arm): Participants receive standard of care therapy.
- Conventional Therapy + Methylene Blue (MB) 0.025%: Participants receive 0.025% dose methylene blue PO to swish and spit for 5 minutes every 6 hours then receive standard of care therapy.
- Conventional Therapy + Methylene Blue (MB) 0.05%: Participants receive 0.05% dose methylene blue PO to swish and spit for 5 minutes every 6 hours then receive standard of care therapy.
- Conventional Therapy + Methylene Blue (MB) 0.1%: Participants receive 0.1% dose methylene blue PO to swish and spit for 5 minutes every 6 hours then receive standard of care therapy.
Period: Overall Study
Arm/Group | Conventional Therapy (Controlled Arm) | Conventional Therapy + Methylene Blue (MB) 0.025% | Conventional Therapy + Methylene Blue (MB) 0.05% | Conventional Therapy + Methylene Blue (MB) 0.1%
Started | 16 | 15 | 14 | 15
Completed | 16 | 15 | 14 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Therapy (Controlled Arm) | Conventional Therapy + Methylene Blue (MB) 0.025% | Conventional Therapy + Methylene Blue (MB) 0.05% | Conventional Therapy + Methylene Blue (MB) 0.1% | Total
Number analyzed (Participants) | 16 | 15 | 14 | 15 | 60
Age, Continuous [Median (Full Range); unit: years] | 48 [26 to 65] | 45 [26 to 76] | 43 [21 to 70] | 32 [19 to 75] | 43 [19 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 5 | 6 | 22
  Male | 10 | 10 | 9 | 9 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 1 | 3
  White | 15 | 11 | 11 | 11 | 48
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 14 | 15 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Scores Assessed Within the Numeric Rating Scale (NRS) Component of the Modified Harris Mucositis-related Pain Assessment Tool
Description: Oral mucositis pain reduction (measured by using the Numeric Rating Scale (NRS); from 0, representing no pain, to 10, representing the worst possible pain) from baseline to 7 days post treatment. The pain scale is included in the Modified Harris mucositis-related pain assessment tool.
Time Frame: Baseline up to day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Therapy (Controlled Arm) | Conventional Therapy + Methylene Blue (MB) 0.025% | Conventional Therapy + Methylene Blue (MB) 0.05% | Conventional Therapy + Methylene Blue (MB) 0.1%
Number analyzed (Participants) | 16 | 15 | 14 | 15
score on a scale | 1.69 (3.09) | 5.2 (2.81) | 4.54 (2.93) | 5.15 (2.64)
Statistical Analysis 1: Comparison: Conventional Therapy (Controlled Arm) vs Conventional Therapy + Methylene Blue (MB) 0.025% vs Conventional Therapy + Methylene Blue (MB) 0.05% vs Conventional Therapy + Methylene Blue (MB) 0.1%; Test type: Other; p = 0.0034, ANOVA

2. Secondary Outcome: Change in Oral Function Burden (OFB) Scores
Description: Oral functioning (eat, swallow, talk: unable=2, difficulty=1, able=0. Oral functioning score is the total score of 3 categories, ranged 0-6). Scale is included in the Modified Harris mucositis-related pain assessment tool. Measurements are obtained at day 0, 1, 2, and 7. Modified Harris mucositis-related pain assessment tool. Lowest value=0 representing normal. Highest value =6 representing worst outcome.
Time Frame: Baseline up to day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Therapy (Controlled Arm) | Conventional Therapy + Methylene Blue (MB) 0.025% | Conventional Therapy + Methylene Blue (MB) 0.05% | Conventional Therapy + Methylene Blue (MB) 0.1%
Number analyzed (Participants) | 16 | 15 | 14 | 15
score on a scale | 0.81 (1.11) | 2.47 (1.55) | 2.79 (1.72) | 2.87 (1.60)
Statistical Analysis 1: Comparison: Conventional Therapy (Controlled Arm) vs Conventional Therapy + Methylene Blue (MB) 0.025% vs Conventional Therapy + Methylene Blue (MB) 0.05% vs Conventional Therapy + Methylene Blue (MB) 0.1%; Test type: Other; p = 0.0008, ANOVA

3. Secondary Outcome: World Health Organization Oral Mucositis Severity Grades
Description: Used the WHO grading system (0= no mucositis, 3=severe mucositis) The clinical severity of the OM was documented only at enrollment point to the study. Most of the patients had the grade 3 mucositis (Soreness/erythema + ulceration + ability to use a liquid diet only), per World Health Organization criteria. See table below which indicates the description of the various grades.
  Grade Description 0 No changes
  1. Soreness/erythema
  2. Soreness/erythema + ulceration + ability to eat solid foods
  3. Soreness/erythema + ulceration + ability to use a liquid diet only
  Secondary endpoint included oral functioning burden (0=normal, 6= worse oral function) (OFB; measured on a scale of 0, representing normal, to 6, meaning total inability, reflecting a total score of three categories: the ability to eat, swallow, and talk, each scored as unable = 2, difficult = 1, able = 0).
Time Frame: Up to day 2
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Therapy (Controlled Arm) | Conventional Therapy + Methylene Blue (MB) 0.025% | Conventional Therapy + Methylene Blue (MB) 0.05% | Conventional Therapy + Methylene Blue (MB) 0.1%
Number analyzed (Participants) | 16 | 15 | 14 | 15
Participants
  Grade 2 | 1 | 0 | 1 | 4
  Grade 3 | 15 | 15 | 13 | 11

4. Secondary Outcome: Morphine Equivalent Daily Doses (MEDD)
Description: Morphine equivalent daily dose (MEDD) used for oral mucositis pain at 2 post MB administration.
  Before the study was implemented, it was observed that many patients had pain resolved just within a few doses. Therefore, the study aimed to cover only 100 cc of MB, which typically last about 2 days. Some patients requested more MB after the two days which had to be provided by the pharmacy and ordered by the primary team and paid by patient insurance. This was considered out of the study, but the patients were still followed. Also, there was no average, only self-reported level of pain from the patient at point of data collection.
Time Frame: Baseline to Day 2
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Conventional Therapy (Controlled Arm) | Conventional Therapy + Methylene Blue (MB) 0.025% | Conventional Therapy + Methylene Blue (MB) 0.05% | Conventional Therapy + Methylene Blue (MB) 0.1%
Number analyzed (Participants) | 16 | 15 | 14 | 15
mg | 117.5 [16.4 to 825] | 115 [12.5 to 535] | 107 [15 to 648] | 120 [5 to 3153]
Statistical Analysis 1: Comparison: Conventional Therapy (Controlled Arm) vs Conventional Therapy + Methylene Blue (MB) 0.025% vs Conventional Therapy + Methylene Blue (MB) 0.05% vs Conventional Therapy + Methylene Blue (MB) 0.1%; Test type: Other; p = 0.9182, Fisher Exact

5. Secondary Outcome: Pain Duration
Description: Measured the days the patient was in pain. The study aimed to cover only 100 cc of MB, which typically last about 2 days. Some patients requested more MB after the two days which had to be provided by the pharmacy and ordered by the primary team and paid by patient insurance. This was considered out of the study, but the patients were still followed. We followed for 30-90 days (no treatment for 30-90 days), only to observe for AEs. Also, there was no average, only self-reported level of pain from the patient at point of data collection.
Time Frame: Up to 30-90 days
Measure: Median (Full Range); unit: days
Arm/Group | Conventional Therapy (Controlled Arm) | Conventional Therapy + Methylene Blue (MB) 0.025% | Conventional Therapy + Methylene Blue (MB) 0.05% | Conventional Therapy + Methylene Blue (MB) 0.1%
Number analyzed (Participants) | 16 | 15 | 14 | 15
days | 5.5 [3 to 8] | 8 [2 to 90] | 6 [1 to 43] | 5 [2 to 30]
Statistical Analysis 1: Comparison: Conventional Therapy (Controlled Arm) vs Conventional Therapy + Methylene Blue (MB) 0.025% vs Conventional Therapy + Methylene Blue (MB) 0.05% vs Conventional Therapy + Methylene Blue (MB) 0.1%; Test type: Other; p = 0.1046, Fisher Exact

ADVERSE EVENTS:
Time Frame: Baseline, Day 0, Day 1, Day 2, Day 7 and Day 30-90
Arm/Group | Conventional Therapy (Controlled Arm) | Conventional Therapy + Methylene Blue (MB) 0.025% | Conventional Therapy + Methylene Blue (MB) 0.05% | Conventional Therapy + Methylene Blue (MB) 0.1%
All-Cause Mortality (participants affected / at risk) | 0/16 | 1/15 | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/14 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT03469284/Prot_SAP_000.pdf